CLINICAL TRIAL: NCT05780359
Title: A Multicenter, Randomized, Controlled, Superiority Clinical Trial to Evaluate the Safety and Efficacy of Drug-eluting Peripheral Arterial Stent System（G-stream） in the Treatment of the Above-the-knee Femoropopliteal Artery Stenosis or Occlusion
Brief Title: Evaluating the Safety and Efficacy of the G-stream® Drug-Eluting Stent in the Above-the-Knee Femoropopliteal Artery
Acronym: G-streamPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP-GS009
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Artery Disease
Keywords: drug eluting stent; drug coating ballon; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug eluting stent (Experimental): Device: Drug-eluting peripheral arterial（G-stream） stent system Manufacturer：Alain Medical (Beijing) Co., Ltd.
  Interventions: Device: Drug eluting stent
- Drug coating balloon (Active Comparator): Device: AcoArt-Orchid® Drug Eluting Balloon Catheter Manufacturer: Acotec Scientific Co., Ltd
  Interventions: Device: drug coating balloon

INTERVENTIONS:
Device: Drug eluting stent — Sirolimus drug-eluting self-expanding stent available from 20mm to 250mm in length, 3.5mm to 7.5mm in diameter of superficial femoral and proximal popliteal arteries (SFA/PPA) cases for inhibiting in-stent restenosis and improve long-term outcome.
  Arms: Drug eluting stent
Device: drug coating balloon — A proprietary lipophilic coating technology that uses magnesium sterate as excipient, facilitates paclitaxel transfer to the vessel wall, enhances drug delivery, and brings minimal downstream effect. Available from 20mm to 300 mm in length, 3mm to 12 mm in diameter, fits every SFA cases, reduces radiation exposure time.
  Other Names: drug eluting percutaneous transluminal angioplasty (PTA) balloon
  Arms: Drug coating balloon

SUMMARY:
A multicenter, randomized, controlled, superiority clinical trial to evaluate the efficacy and safety of drug-eluting peripheral arterial stent system（G-stream） in the treatment of femoropopliteal artery stenosis or occlusion.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of the drug-eluting peripheral arterial stent system（G-stream) in the treatment of superficial femoral artery and/or proximal popliteal artery. Taking the drug eluting balloon catheter (AcoArt-Orchid) as control.

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria：

  1. Age from 18 to 80 years, male or female;
  2. Patients with Lower extremity peripheral artery disease (PAD);
  3. With Rutherford classification between 2 and 5;
  4. Patients understand the purpose of the study, voluntary participation of the study, signs the consent form, willing and able to comply with all requirements, and agrees to attend all required follow-up visits;
* Angiographic Inclusion Criteria： 5.Single lesions or tandem lesions located in the SFA and/or PPA:

  1. Degree of stenosis ≥ 70% and <100%, Total lesion length ≥ 20 mm and ≤ 250 mm; or
  2. Occlusive lesions, total lesion length ≤ 150 mm; or
  3. Series of lesions, total lesion length ≤ 250 mm and length of occlusive lesions ≤ 150 mm; 6.Vessel diameter ≥ 3.5 and ≤ 7.5 mm by visual angiographic assessment; 7.Re-entry device reach and cross a target lesion successfully; 8.Residual stenosis after predilation ≤ 50% without dissection characterized as type D or greater； 9. Patent homolateral iliac inflow (stenosis ≤ 50% ) or homolateral iliac inflow lesion received successfully treated i.e., residual stenosis < 30% after treatment, without severe flow-limiting dissection characterized as type D or greater, without thrombosis, embolism or other serious adverse events; 10.Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (stenosis ≤ 50%) to the ankle or foot before procedure or with planned intervention.

Exclusion Criteria:

-General Exclusion Criteria：

1. Wtih vasculitis or Berger disease;
2. With severe coagulation disorders or uncontrolled severe infections, not suitable for intervention procedure;
3. Known hypersensitivity or contraindication to aspirin, clopidogrel, heparin, paclitaxel, rapamycin, contrast dye or others;
4. History of distal amputation (above the metatarsal) in the target limb or contralateral limb;
5. Severe renal insufficiency (creatinine > 221 umol/L);
6. History of local thrombolysis or systemic thrombolysis within 48 hours prior to procedure;
7. History of acute myocardial infarction within 30 days prior to procedure;
8. History of major surgery（i.e., open cardiac operation, open abdominal surgery or open operation for peripheral artery disease) within 30 days prior to procedure;
9. History of alimentary tract hemorrhage within 3 months prior to procedure;
10. History of stroke/cerebrovascular accident (CVA) within 6 months prior to procedure;
11. Life expectancy <12 months;
12. History of stent, drug-coated balloon or bypass surgery in the target lesion;
13. Use of atherectomy, laser, cryoplasty or other debulking devices in the target lesion during the index procedure;
14. Pregnant, breast feeding, or plan to become pregnant;
15. Current participation in another investigational drug or device clinical study;
16. According to the judgement of the investigator, other situations that are not suitable for enrollment;

    * Angiographic Exclusion Criteria:
17. Heavily calcified lesions;
18. Presence of aneurysm in the target vessel;
19. Acute or subacute thrombosis of the target vessel;
20. History of graft intervention in the target limb.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Reaching Primary patency | 12 months
  Primary patency defined as freedom from clinically-driven target lesion revascularization and CT angiography diagnosis of freedom from restenosis (ie, stenosis ≤ 50%);

SECONDARY OUTCOMES:
Device success rate | During the procedure
  Device success was defined as successful arrival of stent/balloon to the lesion. And subsequent release of the stent delivery system or dilation of balloon. Then withdraw delivery system successfully.
Procedural success rate | During the procedure
  Procedural success was defined as delivery and deployment of the assigned stent/balloon to the target lesion to achieve residual angiographic stenosis no greater than 50% for balloon and 30% for stent.
Clinical success rate | 12 months
  Clinical success was defined as procedural success without server complications (death, target limb major amputation and/or target lesion revascularization (TLR).
Percentage of Participants With TLR and clinical drived-TLR (CD-TLR) | 30 days, 3 months, 6 months and 12 months
  TLR is defined as any surgical or percutaneous intervention to the target lesion(s) after the index procedure.
Percentage of Participants With Target Vessel Revascularization (TVR) and Clinical Drived-TVR (CD-TVR) | 30 days, 3 months, 6 months and 12 months
  TVR is defined as any surgical or percutaneous intervention to the target vessel(s) after the index procedure.
Percentage of Participants With Major Adverse Events (MAEs) | 30 days, 3 months, 6 months and 12 months
  MAEs defined as all-cause death, target limb major amputation and/or target lesion revascularization (TLR).
Percentage of Participants With all-cause Death | 30 days, 3 months, 6 months and 12 months
Distribution of Rutherford classification | 30 days, 3 months, 6 months and 12 months
  Changing in categories of Rutherford classification.
Distribution of Ankle Brachial Index(ABI) | 6 months and 12 months
  Changing in ABI between 6 to 12 months.
Percentage of Participants With Lower Extremity Arterial Thrombosis | 30 days, 3 months, 6 months and 12 months
Percentage of Participants with major and minor amputations of the treated leg | 30 days, 3 months, 6 months and 12 months
  Major amputation defined as amputation above the ankle and minor as below the ankle.

OTHER OUTCOMES:
Adverse Events (AE) and Serious Adverse Events (SAE) related to Device | 24 months
  Percentage of Participants with AE and SAE related to device.
other Adverse Events (AE) and Serious Adverse Events (SAE) | 24 months
  Percentage of Participants with AE and SAE not related to device.
Percentage of Participants Reaching Primary patency | 24 months
  Primary patency defined as freedom from clinically-driven target lesion revascularization and CT angiography diagnosis of freedom from restenosis (ie, stenosis ≤ 50%).
Percentage of Participants With TLR and CD-TLR | 18 months and 24 months
  TLR is defined as any surgical or percutaneous intervention to the target lesion(s) after the index procedure.
Percentage of Participants With TVR and CD-TVR | 18 months and 24 months
  TVR is defined as any surgical or percutaneous intervention to the target vessel(s) after the index procedure.
Percentage of Participants With MAEs | 18 months and 24 months
  MAEs defined as all-cause death, target limb major amputation and/or target lesion revascularization (TLR).
Percentage of Participants With all-cause Death | 18 months and 24 months
Distribution of Rutherford classification | 18 months and 24 months
  Changing in categories of Rutherford classification.
Distribution of Ankle Brachial Index(ABI) | 24 months
  Changing in ABI during 24 months.
Percentage of Participants With Lower Extremity Arterial Thrombosis | 18 months and 24 months
Percentage of Participants with major and minor amputations of the treated leg | 18 months and 24 months
  Major amputation defined as amputation above the ankle and minor as below the ankle.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DOTTER CT, JUDKINS MP. TRANSLUMINAL TREATMENT OF ARTERIOSCLEROTIC OBSTRUCTION. DESCRIPTION OF A NEW TECHNIC AND A PRELIMINARY REPORT OF ITS APPLICATION. Circulation. 1964 Nov;30:654-70. doi: 10.1161/01.cir.30.5.654. No abstract available. PMID 14226164
- [Background] Gruntzig A, Hopff H. [Percutaneous recanalization after chronic arterial occlusion with a new dilator-catheter (modification of the Dotter technique) (author's transl)]. Dtsch Med Wochenschr. 1974 Dec 6;99(49):2502-10, 2511. doi: 10.1055/s-0028-1108161. No abstract available. German. PMID 4434847
- [Background] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Zeller T, Roubin GS, Burket MW, Khatib Y, Snyder SA, Ragheb AO, White JK, Machan LS; Zilver PTX Investigators. Paclitaxel-eluting stents show superiority to balloon angioplasty and bare metal stents in femoropopliteal disease: twelve-month Zilver PTX randomized study results. Circ Cardiovasc Interv. 2011 Oct 1;4(5):495-504. doi: 10.1161/CIRCINTERVENTIONS.111.962324. Epub 2011 Sep 27. PMID 21953370
- [Background] Dake MD, Ansel GM, Jaff MR, Ohki T, Saxon RR, Smouse HB, Machan LS, Snyder SA, O'Leary EE, Ragheb AO, Zeller T; Zilver PTX Investigators. Durable Clinical Effectiveness With Paclitaxel-Eluting Stents in the Femoropopliteal Artery: 5-Year Results of the Zilver PTX Randomized Trial. Circulation. 2016 Apr 12;133(15):1472-83; discussion 1483. doi: 10.1161/CIRCULATIONAHA.115.016900. Epub 2016 Mar 11. PMID 26969758
- [Background] Muller-Hulsbeck S, Keirse K, Zeller T, Schroe H, Diaz-Cartelle J. Twelve-Month Results From the MAJESTIC Trial of the Eluvia Paclitaxel-Eluting Stent for Treatment of Obstructive Femoropopliteal Disease. J Endovasc Ther. 2016 Oct;23(5):701-7. doi: 10.1177/1526602816650206. Epub 2016 May 18. PMID 27193308
- [Background] Muller-Hulsbeck S, Keirse K, Zeller T, Schroe H, Diaz-Cartelle J. Long-Term Results from the MAJESTIC Trial of the Eluvia Paclitaxel-Eluting Stent for Femoropopliteal Treatment: 3-Year Follow-up. Cardiovasc Intervent Radiol. 2017 Dec;40(12):1832-1838. doi: 10.1007/s00270-017-1771-5. Epub 2017 Sep 25. PMID 28948322
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254